CLINICAL TRIAL: NCT04252092
Title: Effects Of Sensory Training and Electrical Stimulation in Sole of The Foot on Proprioceptive and Cortical Sensations in Patients With Acute Hemiplegia
Brief Title: Effects Of Sensory Training and Electrical Stimulation on Sole of The Foot Sensations in Patients With Acute Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: i79zrwdy
Record Dates: First submitted 2019-12-17; First posted 2020-02-05 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Hemiplegia; Stroke, Acute; Sensory Disorders
Keywords: Electrical stimulation; Sensory education; Sensory evaluation; Stroke; Proprioception
MeSH Terms: conditions — Hemiplegia; Stroke; Sensation Disorders | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Group (Experimental): 15 patients who will be applied 15 sessions of sensory training
  Interventions: Other: Sensory training
- Electrical Stimulation Group (Experimental): 15 patients who will be applied 15 sessions of electrical stimulation
  Interventions: Other: Electrical stimulation

INTERVENTIONS:
Other: Sensory training — 15 session,20 minutes sensory training program
  Arms: Sensory Group
Other: Electrical stimulation — 15 session,20 minutes electrical stimulation program
  Arms: Electrical Stimulation Group

SUMMARY:
The aim of this study is to investigate the effects of the sole of foot sensory education and electrical stimulation on proprioceptive and cortical senses in patients with acute hemiplegia.

DETAILED DESCRIPTION:
Hemiplegia is a syndrome characterized by disorders of motor and sensory functions, speech and mental abilities. Hemiplegia is a common neurological problem in the world and is the third most common cause of death.

In addition to motor loss in patients after stroke, sensory problems are accompanied and close to 60% of stroke patients experience sensory problems. In a limited number of studies in the literature, it is stated that sensory impairment in the lower extremity negatively affects standing, walking speed, balance during ambulation and symmetrical gait. At the same time, it has been proven that the sole of the foot sense plays an important role in the balance of sitting, standing up and performing independent daily living activities. After a stroke, sensory training increases functionality, patients with sensory training recover faster, mobility, balance and daily life activities become better, and daily life improvement is expressed. The purpose of sensory training is to maximize the patient's learning through the connection between environment and repetitive activities.

The aim of this study is to compare the effects of neurodevelopmental physiotherapy program combined with sensory training or electrical stimulation on the sole of the foot proprioceptive and cortical senses in individuals diagnosed with hemiplegia.

There is no study on how proprioceptive and cortical sensations will be affected in acute hemiplegic patients if sensory training and electrical stimulation are added to the classical treatment program. By finding and comparing the effects of active (sensory training) and passive treatment (electric stimulation) with this study, it was planned to propose an effective treatment protocol for developing the sole of the foot senses to the experts working in this field.

As a result, purpose of the study is to prevent inadequate sensory input in hemiplegic patients from adversely affecting quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participating to the study in a voluntary basis
* Patients with 50-80 years old
* A stroke diagnosis by a neurologist
* A stroke attack within 6 months
* Minimum 18 points from Mini Mental Test
* Medically stable

Exclusion Criteria:

* Unstable condition
* Other neurological or orthopaedic problems that will affect function other than stroke
* Uncontrolled hypertension
* Diabetic foot ulcers
* Part/total foot amputation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eksen Sağlık, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensory Group | Electrical Stimulation Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensory Group | Electrical Stimulation Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.2) | 69.4 (8.3) | 67.6 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Assessment Of Joint Position Sense
Description: Joint position sense assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. The patient's eyes will be closed. One of the foot on the hemiplegic side of the patient will be brought to a certain position and the patient will be asked to bring the other extremity to a similar position.
  In the case of the correct response to 8 and above from ten attempts, the sense of sensation is considered normal; correct response between 3-7, the sense of sensation is considered decreased; correct response 3 and below, the sense of sensation is considered lost. Higher scores mean better outcomes with 0 being minimum and 10 being maximum.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
correct responses
  Baseline | 5.0 (2.8) | 6.4 (3.0)
  Week 3 | 8.1 (2.3) | 8.6 (2.1)

2. Primary Outcome: Assesment of Joint Passive Motion Sense
Description: Joint passive motion sense assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. The patient's eyes will be closed. One of the patient's big toe in hemiplegic their side will be held on either side and moved up or down. During this time, the patient will be asked to indicate the direction of the movement.
  In the case of the correct response to 8 and above from ten attempts, the sense of sensation is considered normal; correct response between 3-7, the sense of sensation is considered decreased; correct response 3 and below, the sense of sensation is considered lost. Higher scores mean better outcomes with 0 being minimum and 10 being maximum.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
correct responses
  Baseline | 5.3 (2.3) | 6.8 (1.8)
  Week 3 | 8.4 (1.4) | 8.5 (1.3)

3. Primary Outcome: Assessment of Vibration Sense
Description: Vibration sense assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. It is evaluated with a vibrating diapason. While the eyes are closed, the diapason will be placed on the tip of the big toe of the hemiplegic foot, the patient will be asked if the vibration is felt or not. If it is felt, this time the patient will be asked to indicate the moment when the vibration ends. Thus, the time it detects the vibration is determined. This period is about 20 seconds in normal youth. As the age progresses, it should be remembered that vibration time is shortened in lower extremities.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
seconds
  Baseline | 2.5 (2.2) | 4.2 (4.3)
  Week 3 | 6.6 (3.3) | 6.4 (4.5)

4. Primary Outcome: Assesment of Deep Pain Sense
Description: Deep pain sense assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. If the Achilles tendon is squeezed or the muscles are severely suppressed, it is investigated whether or not the pain is felt. If pain is felt, the result will be counted as positive. The positive result is an unwanted result.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: percentage of positive results
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
percentage of positive results
  Baseline | 66.7 (4.5) | 53.3 (4.5)
  Week 3 | 13.3 (3.2) | 6.7 (2.1)

5. Primary Outcome: Assessment of Two-point Discrimination
Description: Two-point discrimination sense assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. The points of the blunt wig will be held against the hemiplegic sole of the foot at different distances from each other. Instruct the client to respond to each touch, by saying one point or two points. Eyes should be closed during the examination. When the patient feels two, it will be noted how far away in cm away from the wig.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
cm
  Baseline | 7.5 (2.6) | 6.9 (2.8)
  Week 3 | 3.1 (1.2) | 3.6 (1.6)

6. Primary Outcome: Assessment of Graphesthesia
Description: Graphesthesia assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. The patient will be asked to estimate a letter or number written the sole of the hemiplegic foot with a blunt object while the eyes are closed.
  In the case of the correct response to 8 and above from ten attempts, the sense of sensation is considered normal; correct response between 3-7, the sense of sensation is considered decreased; correct response 3 and below, the sense of sensation is considered lost. Higher scores mean better outcomes with 0 being minimum and 10 being maximum.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
correct responses
  Baseline | 3.9 (1.9) | 3.1 (1.4)
  Week 3 | 6.8 (1.8) | 5.7 (2.6)

7. Primary Outcome: Assessment of Tactile Localization Sense
Description: Tactile localization sense assessment will be applied to all subjects (30 patients) at the beginning and end of treatments. Patients will be stimulated on 10 different locations of the hemiplegic sole of the foot. They will be asked to localize the touch. The response will be recorded.
  In the case of the correct response to 8 and above from ten attempts, the sense of sensation is considered normal; correct response between 3-7, the sense of sensation is considered decreased; correct response 3 and below, the sense of sensation is considered lost. Higher scores mean better outcomes with 0 being minimum and 10 being maximum.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
correct responses
  Baseline | 6.3 (2.3) | 7.1 (1.9)
  Week 3 | 8.7 (1.5) | 8.8 (1.0)

8. Primary Outcome: Assessment of Tactile Inattention
Description: Tactile inattention assessment will be applied to all subjects (30 patients) at the beginning and end of treatments.The patient will close his eyes. The right and the left half of the body will be needled at the same time. The patient with tactile inattention perceives only one of them which is counted as positive. The positive result is an unwanted result.
Time Frame: Baseline and Week 3
Measure: Mean (Standard Deviation); unit: percentage of positive results
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
percentage of positive results
  Baseline | 60 (6.5) | 26.7 (6.5)
  Week 3 | 20 (2.1) | 13.3 (3.4)

9. Secondary Outcome: Assessment Of Cognitive Level
Description: Mini-mental test will be applied to all subjects (30 patients) at the beginning of treatments. A mini-mental test will be performed to evaluate the patient's cognitive level. This test will be used because it evaluates orientation, recording memory, attention, and computation, remembering and language, orientation, praxis skills.
  In the test consisting of 30 questions and 30 points, a total of ≥25 points were considered normal, 21-24 points Light, 10-20 points medium, and ≤9 serious cognitive disorders. Higher scores mean better outcome with 0 being minimum and 30 being maximum.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensory Group | Electrical Stimulation Group
Number analyzed (Participants) | 15 | 15
score on a scale | 23 (2.9) | 22.9 (4.1)

ADVERSE EVENTS:
Time Frame: 4 Months
Description: No adverse effects has been found as this study is applied on the parts of the body that is not relevant to their vital signs.
Arm/Group | Sensory Group | Electrical Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04252092/SAP_000.pdf
  • Informed Consent Form (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04252092/ICF_001.pdf
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04252092/Prot_002.pdf